CLINICAL TRIAL: NCT00819702
Title: Preventing Child Maltreatment: A Role for Community Pediatricians
Brief Title: A Safe Environment for Every Kid (SEEK): A Model for Primary Care
Acronym: SEEK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HP-00040157 (H-27327); 1R49CE000588 (NIH)
Record Dates: First submitted 2009-01-07; First posted 2009-01-09 (Estimated); Last update posted 2023-05-08 (Actual); Status verified 2019-11

CONDITIONS: Child Maltreatment
Keywords: child abuse prevention; primary care; professional education in primary care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Model Care (Experimental): The Model Care approach was implemented in 7 practices, where PCPs were trained to address major risk factors for CM, including maternal depression, alcohol/substance abuse, intimate partner violence, food insecurity, harsh punishment and major stress. We taught how they can be briefly assessed and initially addressed. The initial training consisted of one 4-hour in-person session. Use of the Parent Screening Questionnaire (PSQ) was discussed, as was the importance of applying it universally during regular checkups. PCPs SEEK Parent Handouts on each targeted problem. We held 1-hour booster sessions every 6 months over the subsequent 2.5 years.
  Interventions: Other: Model Care
- Standard Care (No Intervention): PCPs in Standard Care group served as the controls. They continued to practice as usual.

INTERVENTIONS:
Other: Model Care — The Model Care provided training to pediatric health care providers to assess parental psychosocial risk factors to child maltreatment.
  Arms: Model Care

SUMMARY:
Our broad goal is to help prevent child maltreatment (CM) by modifying pediatric practice to be more responsive to prevalent psychosocial needs of many children and families.Training pediatricians to address key risk factors for CM, the Safe Environment for Every Kid (SEEK) model aims to support parenting and family functioning, reducing the risk for CM while helping promote children's health, development and safety. We are building upon the existing pediatric primary care system and strengthening the training of pediatricians. The project also builds on our extensive research and clinical expertise in CM and in prevention (Black & Dubowitz, 1999, Dubowitz et al., 1998, 1999, in press; Dubowitz & Guterman, 2005, Gaudin & Dubowitz, 1997).

We have developed and implemented an enhanced model of pediatric primary care, taking advantage of the enormous opportunities of the existing pediatric primary care system, with its regular contact with young children and parents (Dubowitz & Newberger, 1989; Dubowitz, 1989, 1990; Green, 1994). Pediatricians typically devote over half their time to checkups, focusing on prevention. There is increasing recognition that pediatric care must incorporate aspects of parental and family functioning and collaborate with community resources (Academy of Pediatrics, 1998; Green, 1994b). The broad goal of this project is to implement concepts that have been embraced by the field of pediatrics, but have not been applied and tested.

DETAILED DESCRIPTION:
The SEEK project, funded by a CDC grant to the Division of Child Protection at the University of Maryland School of Medicine, attempts to offer a comprehensive and practical office-based approach to the identification and assessment of risk factors for child maltreatment, integrated into the delivery of well child health care.

Review of the literature identifies four major risk factors leading to child maltreatment, 1) maternal depression, 2) alcohol and substance abuse, 3) domestic violence, and 4) parental stress and poor coping. The project has several "arms" to address these risk factors. Initially, there is training to help busy primary care providers (PCPs) address the targeted problems in the pediatric office setting. The second phase is the introduction of a brief screening questionnaire into selected well child visits to identify these risk factors in families. If risk factors are present, the PCP will briefly assess the problem. A project social worker is available (by phone or in the office) to help address the problem, and to aid the families in accessing community resources. Another part of the project assesses the validity of the screening questionnaire against several "gold standard" measures used to diagnose the targeted risk problems.

The training focused on the four major factors described. We used realistic office scenarios and offered participants the opportunity to use newly learned management strategies in addressing them. Small group experience with adequate time for processing and practice were utilized. Scheduling was done in conjunction with the participating offices. An advisory committee of practicing community pediatricians and office personnel offered consultation on all phases of the program, as well as strategies to efficiently integrate the program into office practice. The project enlisted 102 PCPs in 18 practices with half serving as controls. Those in the intervention arm received the training. Study health care offices used the one-page SEEK screening questionnaire in their practices. Control pediatricians made no change to their current practice, and continued to provide standard care. Parents were given the questionnaire, in the office, before the 2 and 15 month, and 2, 3, 4, and 5 year well child visits. Questionnaires were completed while the parent waited. Questionnaires were quickly and easily read by the PCPat the visit. Significant issues were briefly assessed and addressed during the visit. The project social worker was available to practices for consultation and for direct intervention with families. "Booster sessions," reviewing the educational and intervention materials were held four times during the 2.5 year study period. PCP knowledge, attitudes, level of comfort and perceived competence regarding the targeted problems were assessed at the beginning and end of the training and at the end of the 2nd and 3rd year.

The central objective of the SEEK project was to examine whether parent functioning was improved by addressing common risk factors for child maltreatment, thus strengthening families and helping prevent maltreatment. A subset of parents in the project practices - intervention and control - were approached to participate in the evaluation of the project. Interest in participating was briefly assessed in the practice. A member of the project team contacted interested parents to fully explain what is involved. Parents who agreed to participate completed a survey (on-line or paper) at three different points. Survey completion took about 60 minutes, for which they were modestly compensated.

In addition, to evaluate the project, members of the project team did a chart review, and directly observed practice behavior. We also asked parents' permission to review Department of Social Services records for possible involvement. All participating pediatricians and practices were invited to share in the conclusions at the end of the project.

The SEEK team hopes that this intervention will be the basis for a new and practical approach to the assessment of serious psychosocial risk factors within the framework of health supervision visits. Ultimately, our hope is that the identification and amelioration of these risk factors will help prevent child maltreatment, and improve the lives of many children and their families. We encourage you to join us in developing an innovative approach to help address psychosocial risk factors in pediatric practice.

ELIGIBILITY:
Inclusion Criteria:

* Mother or mother figure accompanying a child under 6 for a regular checkup.
* Fluent english
* Mother agrees to participate
* Health Care provider is provider at involved practice
* Health Care provider agrees to participate

Exclusion Criteria:

* Mother is already participating through another child
* Mother does not speak english
* Mother declines participation
* Health Care providers practice is not involved in study
* Health Care provider declines

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 905 (Actual)
Dates: Start 2006-05; Primary Completion 2009-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Parent to Child Conflict Tactics Scale | Initial contact, 6 months & 12 months after start of study participation

SECONDARY OUTCOMES:
Department of Human Services, Department of Child Protection records. | Child's birth through March 2009

CONTACTS AND LOCATIONS:
Overall Officials: Howard Dubowitz, MD MS, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, School of Medicine, Baltimore, Maryland, United States